CLINICAL TRIAL: NCT03322111
Title: Assessment of Cyclofusion Capabilities of Normal Subjects and Patients With 3D Dynamic Random-dot Stereograms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cantonal Hospital of St. Gallen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Veit Sturm, Prof. Dr., Cantonal Hospital of St. Gallen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-02118
Record Dates: First submitted 2017-10-06; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Cyclofusion Competence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cyclofusion (Experimental)
  Interventions: Diagnostic Test: measurement of the cyclofusion

INTERVENTIONS:
Diagnostic Test: measurement of the cyclofusion — Measurement of the maximal cyclofusion competence with a dynamic 3-D Random-Dot Landolt-C stimulus

SUMMARY:
With this study the investigator wants measure the individual cyclofusion competence from healthy subjects and patients suffering from Strabismus with a only binocularly visible threedimensional Landolt-C stimulus. For this the participant has to look at a 3-D monitor with shutter glasses. The participant is sitting in 2 meter distance in front of the monitor. On the monitor appears the Landolt-C stimulus as a dynamic Random-Dot Stimulus. As long as the participant can fuse the stimulus he will be able to see the Landolt C-ring threedimensional. The participant is then ask to tell in which direction the notch of the Landolt-C ring points out. Once a critical degree of cyclotorsion is reached the participant will no longer be able to see the Landolt C ring and the individual cyclofusion competence is reached.

ELIGIBILITY:
Inclusion Criteria:

* Visual acuity >0,4; Stereopsis

Exclusion Criteria:

* Visual acuity <0,4; no Stereopsis

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-04-20 (Estimated); Study Completion 2019-04-20 (Estimated)

PRIMARY OUTCOMES:
In- and excyclofusion competence in healthy individuals. Change in In- and excyclofusion competence in patients who need a strabismus surgery before and 6 month after surgery. | Once in healthy individuals. Before and 6 month after a (independent from the study) performed strabismus surgery.
  The maximum in- and maximum excyclofusion competence will be measured with the described test set-up. The results will be documented in degree.